CLINICAL TRIAL: NCT04389606
Title: Follow-up Study of Growth, Safety, and Efficacy of an Infant Formula for Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ByHeart (Industry)
Collaborators: Paidion Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SS-101-Follow-up
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy; Term Infants
Keywords: Infant; Infant Formula; Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Formula (SF) (Experimental): New infant formula for term infants
  Interventions: Other: Study Formula (SF); Other: Comparator Formula (CF)
- Comparator Formula (CF) (Active Comparator): Commercially available infant formula for term infants
  Interventions: Other: Study Formula (SF); Other: Comparator Formula (CF)
- Human Milk Reference Group (No Intervention): Human milk

INTERVENTIONS:
Other: Study Formula (SF) — New infant formula for term infants fed ad lib
  Arms: Comparator Formula (CF); Study Formula (SF)
Other: Comparator Formula (CF) — Commercially available infant formula for term infants fed ad lib
  Arms: Comparator Formula (CF); Study Formula (SF)

SUMMARY:
The purpose of this two-month follow-up study is to continue to follow growth, safety, and other health outcomes of infants fed a new infant formula for term infants or comparator formula. A reference group of human milk-fed infants will also be followed. This study is designed in accordance with Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who enrolled and completed the previous phase of the clinical trial: NCT04218929 "Evaluation of Growth, Safety, and Efficacy of an Infant Formula for Healthy Term Infants"

Exclusion Criteria:

* Subjects who did not enroll in the previous phase of the clinical trial: NCT04218929 "Evaluation of Growth, Safety, and Efficacy of an Infant Formula for Healthy Term Infants"

Ages: 16 Weeks to 19 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Weight Gain Velocity | up to 24 weeks
  G/D

SECONDARY OUTCOMES:
Weight Measures | 20 weeks, 24 weeks
  KG
Length Measures | 20 weeks, 24 weeks
  CM
Length Gain Velocity | 20 weeks, 24 weeks
  CM/D
Head Circumference Measures | 20 weeks, 24 weeks
  CM
Weight for age Z-scores | 20 weeks, 24 weeks
  Weight for age Z-scores compared to World Health Organization (WHO) growth standards
Length for age Z-scores | 20 weeks, 24 weeks
  Length for age Z-scores compared to WHO growth standards
Head circumference for age Z-scores | 20 weeks, 24 weeks
  Head circumference for age Z-scores compared to WHO growth standards
Weight for length Z-scores | 20 weeks, 24 weeks
  Weight for length Z-scores compared to WHO growth standards
72-hr record of formula intake at each study visit | 20 weeks, 24 weeks
  oz/d
Blood concentrations of Interleukin-6 (pg/mL), Interleukin-10 (pg/mL), and tumor necrosis factor-alpha (pg/mL) | 24 weeks
  Concentration
Blood concentrations of amino acids (umol/L) | 24 weeks
  Concentration
Human milk composition (concentrations of proteins, lipids, carbohydrates, vitamins, and minerals | 24 weeks
  Concentration
Medically-diagnosed adverse events collected throughout the study period | 16-24 weeks
  Frequency
Parent rating of infant stool consistency at each study visit | 20 weeks, 24 weeks
  Mean. Quinlan et al Likert scale; 0=no bowel movement, 1=hard [dry hard pellets], 2=formed [definite shape, not dry], 3=soft [no definite shape, pasty], 4=loose [no shape, some water], 5=watery [no shape, mainly water]).
Parent report of infant stool frequency at each study visit | 20 weeks, 24 weeks
  Mean
Parent report of infant disposition (fussiness, crying, gas, spit up, Infant Characteristics Questionnaire) at each study visit | 20 weeks, 24 weeks
  Mean
Stool microbiome | 24 weeks
  Fecal microbial taxa and community abundance
Stool metabolome | 24 weeks
  Targeted and Untargeted Metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Devon Kuehn, MD, Study Director — ByHeart, Inc.
Locations (27):
- United States (27):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Watching Over Mothers and Babies, Tucson, Arizona
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - San Gabriel Women's Health, Arcadia, California
  - Northern California Research, Sacramento, California
  - Optum, Colorado Springs, Colorado
  - Topaz Clinical Research, Apopka, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Avanza Medical Research, Pensacola, Florida
  - PAS-Research, Tampa, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Southern Clinical Research, Zachary, Louisiana
  - Sierra Clinical Research, Las Vegas, Nevada
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Schear Family Practice, Dayton, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Institute of Clinical Research, Mentor, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatric Associates, Summerville, South Carolina
  - HMG Primary Care at Sapling Grove, Bristol, Tennessee
  - Jackson Clinic North, Jackson, Tennessee
  - HMG Pediatrics at Kingsport, Kingsport, Tennessee
  - Houston Clinical Research Associates, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - ACRC Trials Plano Pediatrics, Plano, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuehn D, Zeisel SH, Orenstein DF, German JB, Field CJ, Teerdhala S, Knezevic A, Patil S, Donovan SM, Lonnerdal B. Effects of a Novel High-Quality Protein Infant Formula on Energetic Efficiency and Tolerance: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2022 Oct 1;75(4):521-528. doi: 10.1097/MPG.0000000000003490. Epub 2022 Jun 6. PMID 35666855